CLINICAL TRIAL: NCT04241588
Title: Assessment of Neural and Motor Performance in Upper Limb Deficient Subjects Using Discrete and Continuous Tasks. Anatomical Differences of Brain Gray and White Matter Resulting From Unilateral Congenital Upper Limb Loss
Brief Title: Assessment of Neural and Motor Performance
Status: Withdrawn | Type: Observational
Why Stopped: We did not received funding for this project, so we could not initiate enrollment.
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0589-19-FB
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Amniotic Band Syndrome; Upper Extremity Deformities, Congenital
MeSH Terms: conditions — Amniotic Band Syndrome; Upper Extremity Deformities, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- 3D prostheses users: Children with unilateral congenital upper-limb reductions
  Interventions: Device: 3D Printed Upper-limb Prosthesis
- Typically Developing Children: Age- and sex-matched control group of typically developing children.
  Interventions: Other: Control

INTERVENTIONS:
Device: 3D Printed Upper-limb Prosthesis — The fingers and thumb were made of polylactic acid polymer manufactured using industrial 3D printers. The palm, socket, forearm brace, and leveraging the structure were made of polylactic acid which has properties similar to thermoplastic that facilitate post-manufacturing adjustments. Elastic cords placed inside the dorsal aspect of the fingers provided passive finger extension. Finger flexion was driven by non-elastic cords along the palmar surface of each finger and was activated through 20-30 degrees of wrist or elbow flexion. The device will be given to participants so that they may practice using the device at home.
  Other Names: Prosthesis use
  Groups: 3D prostheses users
Other: Control — A 3D printed hand with be fitted to simulate a prosthesis.
  Groups: Typically Developing Children

SUMMARY:
The neural basis underlying motor performance in children using a prosthesis has been severely understudied resulting in minimal empirical evidence. With the use of low-cost 3D printed prosthetics, the purpose of this study is to examine the assessment of primary motor cortex activation and the representation of gray and white matter in a child with congenital limb loss. This will be accomplished by cross-examining results from fNIR and Anatomical Magnetic Resonance Imaging (MRI). The proposed research uses anatomical MRI to test if children with unilateral congenital partial hand reductions demonstrate less gray and white matter in the motor representation zones. Moreover, the proposed research will focus on an assessment of motor performance using continuous and discrete tasks with a robotic manipulandum. Assessment of motor performance and neural networking are critical to increasing our limited knowledge of how the child increases the number of motor repertoires.

DETAILED DESCRIPTION:
The investigators anticipate enrolling a total of 40children between 3 and 18 years of age. Specifically, two groups of children will be recruited; children with unilateral congenital upper-limb reductions (n=20) and age and sex-matched control group of typically developing children (n=20). Considering the effect size from preliminary data and to account for a 10% drop-out rate, a total sample of 40 subjects will provide 80% power to detect a true standardized effect size.

All subjects including controls will attend four data collection sessions that will include: one fitting session, second to obtain a baseline, the third visit will be one month after baseline, and the final visit will be four months after baseline. Participants will attend an initial measurement session to take a 3D scan of the affected and nonaffected upper limbs as well as several anthropometric measurements. During this session, three pictures of the upper limbs will be taken which will also be used to verify the fit the prostheses in a process previously validated by our research team. The subjects will then perform an anatomical MRI scan. The MRI scan is not a clinical scan intended for diagnostic or therapeutic purposes. The research participants will then be asked to come for two testing visits. During the first testing visit (visit 1), participants will be fitted with the prosthesis and required adjustments to improve comfort and avoid pressure point will be performed. After fitting the prosthesis, participants will be given 15 minutes to explore the prosthesis and adjust the tensioner dial to regulate the opening of the fingers to perform the Box and Block Test. After the training and accommodation period, participants will be asked to perform 3 trials of flexion and extension of each wrist with and without the prosthesis and 3 different trials of the Box and Blocks Test for each hand while monitoring neural activity of the primary motor cortex using a fNIRS device. After a brief period of rest and encouragement, the subject will be asked to perform eight trials of discrete (four trials) and continuous (four trials) tasks using a robotic manipulandum (InMotion Arm Robot, Interactive Motion Technologies, Inc., Cambridge, MA, USA). These tasks have been previously used for the assessment of changes in upper-limb performance and the effect of different treatments in the recovering of motor function of children with acquired or congenital hemiparesis, ataxia, and hemiparesis. This data collection performed at baseline will be performed again one and four months after baseline. Eight weeks after the baseline measurements, participants will be asked to visit our laboratory for a second time and perform the same assessments. Between the testing visits, participants will be encouraged to use the prosthesis for a minimum of 2 hours a day.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-80 years.
* Individuals missing any digits, hand, arm, shoulder.
* Any dysfunction of the upper limbs.

Exclusion Criteria:

* Participants who are outside of age range.
* Participants with upper extremity injury within the past month.
* Medical conditions which would be contraindications to wear a prosthetic or assistive device, Such as skin abrasions and musculoskeletal injuries in the upper limbs.

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Nebraska residents and residents from other states will be invited to participate in the research study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Change of mean values of brain hemodynamic responses | Change from baseline of mean values of brain hemodynamic responses at 4 month.
  The oxy-hemoglobin (HbO) and deoxy-hemoglobin (HbR) are two major chromospheres in the blood which absorb NIR light. The concentration of HbO and HbR varies in the capillary blood during the rest and task sessions. Thus, brain functional information can be revealed by the estimation of HbO and HbR. HbT is the total hemoglobin.
Change of hemispheric dominance | Change from baseline of hemispheric dominance at 4 months.
  Measured using the Laterality Index revealing hemispheric dominance. The Laterality index will reveal hemispheric dominance using the following formula:
  Laterality index=(Oxy l-Oxy r)/(Oxy l+Oxy r) In this equation, l represents the channels from the left hemisphere and r indicates the channels from the right hemisphere. The Laterality index value will reveal which channels in the group showed a higher change during the task. Positive values indicate left-hemisphere dominant activation, while negative values indicate a right-hemisphere dominant activation.
Change of synchrony of hand movement | Change from baseline of retention and transfer of motor skills in 4 months.
  The synchrony of hands movement will be quantified as the absolute temporal difference between hands (non-affected hand and affected hand with prosthesis) at six points in time while moving a bilateral instrumented tray.
Change of movement duration | Change from baseline of movement duration at 4 months.
  Movement duration for continuous and discrete tasks will be measured while completing robotic manipulandum tasks.

SECONDARY OUTCOMES:
Satisfaction assessed by the Project-Prosthesis Satisfaction Inventory (CAPP-PSI). | After 1,2, and 4 months
  The parents of the participants select a response for each question using the following categories which are scored from 0 to 4: "not at all" =0, "a little" =1, "somewhat" =2, "a lot" =3, or "very much" =4. A higher score indicates higher satisfaction. The CAPP-PSI is a standardized measure of prosthesis satisfaction in children with limb deficiency.
Satisfaction assessed by the Orthotics Prosthetics Users' Survey (OPUS). | After 1,2, and 4 months
  The parents of the participants select a response for each question using the following categories which are scored from 5=Very Satisfied, 4= Somewhat satisfied, 3=Neither, satisfied nor dissatisfied, 2=Somewhat dissatisfied, 1=Very Dissatisfied. A higher score indicates higher satisfaction. The OPUS is a self-report questionnaire consisting of five modules. Module 5 (OPUS Satisfaction) will be used to assess different satisfaction element.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge M Zuniga, PhD, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: No
Unidentified data